CLINICAL TRIAL: NCT04250623
Title: Dermatological Assessment of Photoallergy and Phototoxicity Under Controlled and Maximised Conditions.
Brief Title: Dermatological Assessment of Photoallergy and Phototoxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: All-S-FA-FT-SO-PAD-074832
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact | interventions — Gels

STUDY DESIGN:
Intervention Model Description: Clinical trial, single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subjects, 18-70 y, healthy (Experimental): subjects, 18-70 y, healthy
  Interventions: Other: Health care product (gel)

INTERVENTIONS:
Other: Health care product (gel) — hyaluronic acid intimate moisturizing gel (to be applied on the subject's skin)

SUMMARY:
This is a clinical study for health care product safety assessment. The research will be conducted with 40 subjects*, aged 18 to 70 years. The product will be applied on the right and/or left participant back for 3 consecutive weeks. After 10 days, will have another application of the same product, which will be removed in 24 hours. Medical evaluation will be available throughout the study to assess possible adverse events.

The objective of the study is to observe the effects of the application of the product on the skin and prove the absence of photoallergy and phototoxicity.

* 29 completed the trial

DETAILED DESCRIPTION:
40 subjects, aged 18 to 70 years, phototypes II to III (according to Fitzpatrick classification). The patch test will be used to verify the absence of photoallergy and phototoxicity by the investigational products. The products will be applied twice a week for 3 consecutive weeks, as they are over semi-occlusive dressings. The product will remain in contact with the skin for 24 hours, after product removal the area will be irradiated with ultraviolet lamp A and B (UVA/UVB). Then, the procedure will be repeated after 10 days of wash out.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to comply with safety guidelines to minimize the risk of contamination to COVID-19;
* Agreement to perform a molecular test for the detection of COVID-19 to enter the study;
* Healthy participants;
* Non-injured skin in the test region;
* Agreement to adhere to the test procedures and requirements and to attend the institute on the day(s) and at the time(s) determined for the evaluations;
* Ability to consent to participation in the study;
* Age from 18 to 70 years;
* Phototype (Fitzpatrick): II and III;
* Any gender

Exclusion Criteria:

* Participants who belong to the risk group for COVID-19, that is, with diabetes, with chronic cardiovascular, renal and respiratory problems, immunosuppressed or other conditions that the physician deems as belonging to the risk group;
* Skin marks in the experimental area;
* Active dermatoses (local or widespread);
* Pregnant or breastfeeding women;
* History of allergic reactions, irritation or intense feelings of discomfort to topical products;
* History of phototoxic or photoallergic reactions;
* History of allergy to materials used in the study;
* History of atopy;
* Personal or family pathological history of skin cancer;
* History of pathologies aggravated or triggered by ultraviolet radiation;
* Carriers of immunodeficiencies;
* Intense sun exposure or tanning session up to 15 days before the initial evaluation;
* Predicted intense sun exposure or tanning session during the course of the study;
* Predicted bathing in the sea, pool or bathtub during the study;
* Participants who practice water sports;
* Dermography;
* Use of the following topical or systemic drugs: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs and corticoids up to 2 weeks prior to selection or, considering deposit corticoids, the interval shall be 1 month prior to selection;
* Use of topical or systemic photosensitizing drugs;
* Treatment with acid vitamin A and/or its derivatives via oral or topical until 1 month before the beginning of the study;
* Aesthetic and/or body dermatological treatment until 3 weeks before selection;
* Vaccination during the study or until 3 weeks before the study;
* Being or having participated in another clinical trial terminated less than 7 days before selection, in case the previous trial is acceptable in use;
* Being or having participated in another clinical trial terminated less than 21 days ago, in case the previous trial is compatible or Adverse Reaction investigative;
* History of absence of adherence or unwillingness to adhere to the study protocol;
* Professionals directly involved in the execution of this protocol and their relatives.
* Participants who have COVID-19, or who present symptoms indicative of the disease in the last 14 days.
* Any condition not mentioned above that, in the opinion of the investigator, may compromise the evaluation of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Absence | 6 weeks
  Absence occurence of phototoxicity and photoallergy

CONTACTS AND LOCATIONS:
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil